CLINICAL TRIAL: NCT03017755
Title: Your Scoliosis Journey: A Survey for Patients Treated for Scoliosis and Their Families
Brief Title: Scoliosis Survey to Development Treatment Decision Tool
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Todd A. Milbrandt, M.D., MD, Mayo Clinic
Other Study IDs: 16-008212
Record Dates: First submitted 2017-01-09; First posted 2017-01-11 (Estimated); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Scoliosis; Adolescence
MeSH Terms: conditions — Scoliosis | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Survey for Patients Treated for Scoliosis and ther Families — Your Scoliosis Journey: A Survey for Patients Treated for Scoliosis and ther Families

SUMMARY:
This is a survey to help understand the influences related to the decision for Adolescent Idiopathic Scoliosis treatment (observation vs. bracing vs. surgery). The investigator then plans to create a decision aid to help families when making a decision about the treatment choice being presented to them.

DETAILED DESCRIPTION:
This survey is designed to help understand the factors that families consider to help make treatment decisions related to Adolescent Idiopathic Scoliosis (AIS). The surveys will then be used to help create a shared decision making tool to help families better understand the treatment options and optimize clinical conversations surrounding AIS treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subject (and/or parent of subject) who has previously been treated for Adolescent Idiopathic Scoliosis (AIS)

Exclusion Criteria:

* Age less than or equal to 12 years

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adolecent Idiopathic Scoliosis (AIS) patients and their families
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2017-04-11 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Number of subjects who completed the survey | Baseline, approximately 3 years
  Number of subjects who completed the survey

CONTACTS AND LOCATIONS:
Overall Officials: Todd A Milbrandt, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials